CLINICAL TRIAL: NCT03620383
Title: Radial Artery Vasodilation With Distal Topical Heat Study
Brief Title: Radial Artery Vasodilation Heat Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ramsey Al-Hakim, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00018794
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-08

CONDITIONS: Radial Artery
Keywords: Transradial access; Radial artery; Vasodilation; Heat
MeSH Terms: conditions — Aneurysm | interventions — Hot Temperature

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat (Experimental): Distal topical heat application
  Interventions: Procedure: Topical Heat
- No Heat (No Intervention): Inactive heat pack to blind the investigator.

INTERVENTIONS:
Procedure: Topical Heat — Warm heat pack applied topically in participant hand.
  Arms: Heat

SUMMARY:
The purpose of this study is to collect data about the efficacy of utilizing distal topical heat application for dilatation of the radial artery. Transradial arterial access is widely accepted as the standard of care for cardiac catheterization procedures due to its increased patient comfort and significantly decreased risk of major vascular complications, and has been recently utilized in increasing volume by the interventional radiology community throughout the world. Due to the small size of the radial artery, catheterization may sometimes be technically difficult. Pre-procedure dilatation can make catheterization significantly easier, and studies have demonstrated the successful ability to dilate the radial artery with the use of topical nitroglycerin and lidocaine. However, the investigators hypothesize that utilizing topical heat applied distally can create a physiologic vasodilatation similar to that created with nitroglycerin and lidocaine, but at a significantly lower cost and with less risk due to no need for application of a medication which has a systemic effect with known side effects. The purpose of this study is to test the efficacy of radial artery vasodilatation with distal topical heat application.

DETAILED DESCRIPTION:
The study will be designed to detect a significant increase in the radial artery diameter of healthy volunteers after the application of a warm heat pack in the palmar aspect of the hand compared to a control group without heat applied to the hand. Employees and students at OHSU will be considered for enrollment as volunteers for this minimal risk study. Informed consent will be obtained from healthy volunteers prior to enrollment. After enrollment, the healthy volunteers will be randomly assigned in a 2:1 ratio to the heat group (Group 1) or the control group (Group 2), respectively. A brief medical history will be obtained from all volunteers, including age, sex, medications, prior interventions, prior surgeries, previous medical diagnoses, allergies, and any history of prior transradial procedures. For protection of confidential health information, brief medical history will be obtained in a private area. The volunteers will then be seated and the left hand placed supinated in a comfortable position on a table. A limited ultrasound of the left radial artery will be performed using grayscale ultrasound. A skin mark will be made with a marker to identify the measurement site. All volunteers will then be given a commercially available warm heat pack and asked to hold gently in their left hand. For the control group (Group 2), the warm heat pack will not be activated. For the heat group (Group 1), the warm heat back will be activated prior to placing in the volunteer's hand. Two investigators will be present. One investigator will be measuring radial artery diameter and will not be aware if the heat pack is activated. The second investigator will be aware of the volunteer's randomly assigned group and will activate the heat pack for the volunteer if they are assigned to Group 1. Over a period of 20 minutes, repeat ultrasound of the left radial artery will be performed in 5 minute intervals.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who are 18-99 years old

Exclusion Criteria:

* Prior left transradial access for procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Al-Hakim, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heat | No Heat
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heat | No Heat | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.4) | 34.2 (9.3) | 36.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 5 | 28
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline radial artery cross sectional area [Mean (Standard Deviation); unit: mm^2] | 2.5 (0.8) | 3.2 (1.1) | 2.7 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Radial Artery Cross Sectional Area
Description: Radial artery cross sectional area after 20 minutes with or without heat application
Time Frame: 20 minutes after application of topical heat
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Heat | No Heat
Number analyzed (Participants) | 30 | 15
mm^2 | 3.4 (1.3) | 3.0 (1.2)

ADVERSE EVENTS:
Time Frame: Day of radial artery measurement
Arm/Group | Heat | No Heat
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 0/30 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03620383/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT03620383/SAP_001.pdf